CLINICAL TRIAL: NCT00291239
Title: Phase 4 Study on the Effect of Partial Sleep Deprivation on Cognition and the IL-6-gp130-System in Individuals With Major Depression
Brief Title: Effect of Partial Sleep Deprivation on Cognition and Cytokines in Individuals With Major Depression
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Zentrum für Integrative Psychiatrie (Other)
Collaborators: German Research Foundation (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: WADE; DFG-SFB 654, C5 "IL-6-MDE"
Record Dates: First submitted 2006-02-09; First posted 2006-02-13 (Estimated); Last update posted 2009-04-03 (Estimated); Status verified 2009-04

CONDITIONS: Major Depression
MeSH Terms: conditions — Depressive Disorder, Major

INTERVENTIONS:
Behavioral: partial sleep deprivation

SUMMARY:
40 patients with the diagnosis of major depression are included. There are two interventions: partial sleep deprivation (PSD) and normal night sleep (CTRL). Patients are randomly assigned to PSD-(2 undisturbed nights)-CTRL or CTRL-(2 undisturbed nights)-PSD. Cytokine-status, neuropsychological and psychopathometric status are assessed pre and post each interventional and control condition.

ELIGIBILITY:
Inclusion Criteria:

* Major depression
* Informed consent

Exclusion Criteria:

* Known epilepsy or previous unexplained loss of consciousness after sleep deprivation
* Bipolar disorder
* Acute or chronic inflammatory diseases
* Psychosis
* Suicidal tendency
* Pregnancy or nursing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2006-02; Primary Completion 2008-12 (Actual); Study Completion 2009-07 (Estimated)

PRIMARY OUTCOMES:
cognition
cytokine concentration

SECONDARY OUTCOMES:
clinical improvement

CONTACTS AND LOCATIONS:
Overall Officials: Dunja Hinze-Selch, MD, Principal Investigator — Zentrum für Integrative Psychiatrie
Locations (1):
- Zentrum für Integrative Psychiatrie, Kiel, Germany